CLINICAL TRIAL: NCT06074224
Title: Sleep Assessment: The Benefits of Identifying Sleep Disturbance Using a Sleep Questionnaire
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, David Ring, Professor of Surgery and Perioperative Care Department, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2020-05-0067
Record Dates: First submitted 2023-09-28; First posted 2023-10-10 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Sleep Disturbance
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinician with Scores (Experimental): The patients in the intervention group will include those for whom their clinician was given their sleep questionnaire result before the visit.
  Interventions: Other: Sleep assessment score
- Clinician without Scores (Active Comparator): The control group will include patients whose clinicians do not view the results, simulating usual care.
  Interventions: Other: No Score

INTERVENTIONS:
Other: Sleep assessment score — The patients in the intervention group will include those for whom their clinician was given their sleep questionnaire result before the visit.
  Arms: Clinician with Scores
Other: No Score — The patients in the control group will include those for whom their clinician was not given their sleep questionnaire result before the visit.
  Arms: Clinician without Scores

SUMMARY:
The investigators are interested in measuring the influence of addressing sleep in the orthopedic setting. This includes assessing patient experience measures (satisfaction with the visit, perceived empathy, communication effectiveness) as well as greater engagement in their healthcare (patient activation). The investigators will also see what factors might be associated with sleep disturbance and if addressing sleep leads to an intervention such as cognitive behavioral therapy.

DETAILED DESCRIPTION:
All adult (18+ years old) new patients seeing a musculoskeletal specialist will be invited to enroll. For the purposes of this trial, The investigators will include people with lesser degrees of sleep disturbance including anyone with a score greater than 3. For people that are enrolled in the trial, the researcher will record the PSQI score and enter at the first page of survey filled out by the patient after meeting. P The patients in the intervention group will include those for whom their clinician was given their sleep questionnaire result before the visit. The control group will include patients whose clinicians do not view the results, simulating usual care. Patients in both groups will fill out a survey entailing demographics, sleep quality, JSPPPE.

ELIGIBILITY:
Inclusion criteria:

1. Adult patients (18+)
2. Orthopedic new visit
3. Sleep disturbance score > 3

Exclusion criteria:

1. Inability to read.
2. Diminished cognition preventing completion of the questionnaires.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Jefferson Scale of Patient's Perceptions of Physician Empathy | through study completion, an average of 6 months
  The Jefferson Scale of Patient's Perceptions of Physician Empathy includes five 7-point scale questions and higher scores indicated greater perceived clinician empathy.

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD, Principal Investigator — Professor of orthopedic surgery at The university of Texas at Austin
Locations (2):
- United States (2):
  - University of Texas Health Austin (UTHA), Austin, Texas
  - University of Texas Health Austin, Austin, Texas

IPD SHARING:
Plan to Share IPD: No